CLINICAL TRIAL: NCT05812131
Title: Web-Based Provider Training for Concurrent Treatment of PTSD and Substance Use Disorders Using Prolonged Exposure (COPEWeb)
Brief Title: COPEWeb Training for Providers
Acronym: COPEWeb
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Medical University of South Carolina (Other); National Center for PTSD (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 21-005
Record Dates: First submitted 2023-03-13; First posted 2023-04-13 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: PTSD; Substance Use Disorders
Keywords: PTSD; substance use disorders; training; providers
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Providers will be randomly assigned to COPEWeb online training or in-person COPE training
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- COPEWEb (Experimental): online COPEWeb training
  Interventions: Behavioral: COPEWeb online training
- COPE In person (Active Comparator): COPE training delivered in person
  Interventions: Behavioral: COPE In Person

INTERVENTIONS:
Behavioral: COPEWeb online training — COPE training delivered via online COPEWEb to providers
  Arms: COPEWEb
Behavioral: COPE In Person — COPE training provided in person to providers
  Arms: COPE In person

SUMMARY:
PTSD and substance use disorders (SUD) are two of the most common and debilitating mental health conditions afflicting military Veterans. PTSD and SUD frequently co-occur and are associated with poorer treatment outcomes. The investigators' team developed a trauma-focused intervention, Concurrent Treatment of PTSD and Substance Use Disorders Using Prolonged Exposure (COPE), which is identified by the VA as a gold standard of behavioral healthcare and was designated as a first-line treatment in the 2025 APA Clinical Practice Guideline for PTSD. However, a critical barrier to ensuring that Veterans with co-occurring PTSD/SUD receive evidence-based treatment is a lack of provider training. This project directly addresses this critical gap by developing a new web-based training program for providers (COPEWeb).

DETAILED DESCRIPTION:
Background: PTSD is the most common mental health disorder among Veterans seeking treatment at Veterans Affairs (VA) hospitals, and more than half of Veterans with PTSD also meet criteria for a substance use disorder (SUD). To address the critical need for PTSD/SUD treatment, members of the investigative team developed Concurrent Treatment of PTSD and Substance Use Disorders Using Prolonged Exposure (COPE), an evidence-based, integrated, trauma-focused treatment identified by the VA as a gold standard of behavioral healthcare. Randomized controlled trials among Veterans demonstrate COPE's efficacy in significantly reducing PTSD and substance use. The majority of Veterans with PTSD/SUD prefer integrated treatment. Significance/Impact: At present, there is a critical shortage of clinicians trained to deliver COPE. Traditional in-person workshops are inefficient and costly. A poll of VA PTSD/SUD Specialists across the country found that 96.9% are interested in receiving COPE training and 99.1% would use a web-based training for COPE if available. A web-based resource for providers is ideal, as it can be rapidly disseminated, is easily accessible, and provides a significant amount of information in a standardized way. This project will directly address this critical gap in provider training to improve the care of Veterans with comorbid PTSD/SUD, enhance treatment delivery using innovative in-session provider assistance tools, and enhance knowledge of cost-benefit of technology-enhanced training. COPEWeb may be particularly useful for providers in rural clinic settings where mental health training is less accessible. This proposal has the potential for high military relevance and an immediate impact on dissemination and uptake of COPE, as well as a long-term impact on the overall health of the millions of Veterans suffering from co-occurring PTSD/SUD. Innovation: A new web-based provider training for COPE will be developed along with a highly innovative provider assistance toolkit to guide clinicians in real-time during sessions to enhance delivery and fidelity to the protocol and reduce provider burden. A panel of national VA experts and dissemination leaders will develop a best practice VA dissemination guideline on disseminating web-based provider trainings. The proposed project has the potential to significantly enhance provider training and increase patient access to evidence-based care. Furthermore, COPEWeb has the potential to serve a novel role in disaster planning to ensure mental health care providers are equipped to address the anticipated post-pandemic needs of Veterans given the rise in post-traumatic stress and alcohol/drug use during the pandemic. Specific Aims: This project aims to 1) develop a new web-based training protocol and innovative delivery aid system to strengthen providers' delivery of COPE to treat Veterans with PTSD/SUD with a high level of fidelity and competence, and 2) compare the COPEWeb training to in-person training on measures of knowledge, satisfaction, and behavior (i.e., fidelity). The cost effectiveness of web-based vs. in-person training will be examined. Methodology: The proposed methods and timeline for the development of COPEWeb are based on the team's prior success developing other widely-used provider training protocols (e.g., PEWeb, CBTIWeb). COPEWeb will be built and refined over the course of three strategic phases: content development, alpha-testing, and beta-testing. Following beta testing, the investigators will compare COPEWeb to in-person training among clinicians. Ongoing assessment will obtain qualitative and quantitative data on measures of provider satisfaction, knowledge, and behavior. Implementation/Next Steps: In collaboration with the investigators' operations partners, VA leadership, and EBP Coordinators, COPEWeb will be rapidly disseminated to mental health providers to increase adoption of evidence-based treatment for PTSD/SUD and improve the quality of mental health care for Veterans and the nation.

ELIGIBILITY:
Inclusion Criteria:

* currently a provider in a behavioral health field (e.g., psychology, psychiatry, counseling)
* at least 18 years old
* English speaking
* able to consistently obtain reliable internet access
* willing to attend a 2-day "live" in-person (or virtual) COPE training if randomly assigned to that condition
* willing to engage in a standardized patient assessment after training
* has no prior formal training in the COPE therapy

Exclusion Criteria:

* received prior training in COPE
* not a provider in the behavioral health field
* non-English speaking
* lack of reliable internet access
* younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-04-05 (Estimated)

PRIMARY OUTCOMES:
IBM Computer Usability Satisfaction Questionnaires (CSUQ) | Through study completion, an average of 8 weeks
  The CSUQ is a 19-item Likert-type (7-point [strongly agree to strongly disagree]) questionnaire that provides an overall usability satisfaction score along with subscales that measure program usefulness, information quality, and interface quality. The CSUQ measure and subscales have good reliability, sensitivity, and validity.
COPE Knowledge Acquisition Test (CKAT) | Change from baseline to study completion, an average of 8 weeks
  The CKAT will be completed at pre- and post-training. The 20-item measure will be scored and the percent of items answered correctly (rated from 0 to 100% correct) will be assessed. Higher scores represent greater knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Sudie E. Back, PhD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No